CLINICAL TRIAL: NCT03873948
Title: Analysis of Serum and Salivary ADMA-Arginine Levels in Patients With Periodontal and Cardiovascular Diseases
Brief Title: Evaluation of Arginine in Periodontal and Cardiovascular Disease
Status: Completed | Type: Observational
Sponsor: University of Messina (Other)
Responsible Party: Principal Investigator, Gaetano Isola, DDS, PhD, Junior Assistant Professor, University of Messina
Other Study IDs: 12-16
Record Dates: First submitted 2019-03-09; First posted 2019-03-14 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Metabolic Disorder; Arginine; Hyperaminoaciduria
MeSH Terms: conditions — Metabolic Diseases; Amino Acid Metabolism, Inborn Errors

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Control: Healthy patients
  Interventions: Other: Evaluation of arginine serum level
- Periodontitis: Patients with periodontal disease
  Interventions: Other: Evaluation of arginine serum level
- Cardiovascular: Patients with cardiovascular disease
  Interventions: Other: Evaluation of arginine serum level
- Periodontitis+Cardiovascular: Patients with both periodontal and cardiovascular disease
  Interventions: Other: Evaluation of arginine serum level

INTERVENTIONS:
Other: Evaluation of arginine serum level — correlation of serum arginine level with periodontal and cardiovascular disease

SUMMARY:
Asymmetric dimethylarginine (ADMA) plays a key role in endothelial function and may be a link for the known interaction of periodontitis and coronary heart disease (CHD). The investigators compared the impact of gingival health, periodontitis (CP), CHD or of both diseases (CP+CHD) on saliva and serum ADMA levels.

DETAILED DESCRIPTION:
The aim of this study was to evaluate a possible association between both saliva and serum ADMA levels in patients with CP and with CHD and if the serum ADMA levels are mediated by serum CRP.

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least 16 teeth
* CP with a minimum of 40% of sites with a clinical attachment level (CAL) ≥2mm and probing depth (PD) ≥4mm;
* Presence of at least ≥2 mm of crestal alveolar bone loss verified on digital periapical radiographs
* Presence of ≥40% sites with bleeding on probing (BOP)

Exclusion Criteria:

* Intake of contraceptives
* Intake of immunosuppressive or anti-inflammatory drugs throughout the last three months prior to the study
* Status of pregnancy or lactation
* Previous history of excessive drinking
* Allergy to local anaesthetic
* Intake of drugs that may potentially determine gingival hyperplasia such as Hydantoin, Nifedipine, Cyclosporin A or similar drugs.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Thus, for this study, 35 patients with CP, 36 patients with CHD, 35 patients with CP+CHD, and 35 healthy subjects will finally enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2014-01-06 (Actual); Primary Completion 2018-08-08 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Clinical Attachment level | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- University of Messina, Messina, Italy

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: 10 years at least